CLINICAL TRIAL: NCT05456581
Title: New Methods to Quantify and Train Eye Movement Strategies in Macular Degeneration
Brief Title: Scotoma Perimetry Oculomotor Training
Acronym: SPOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University of California, Riverside (Other)
Responsible Party: Principal Investigator, Kristina M Visscher, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 300006197 (R21)
Record Dates: First submitted 2022-07-07; First posted 2022-07-13 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Macular Degeneration; Central Visual Impairment
Keywords: plasticity; central vision loss
MeSH Terms: conditions — Macular Degeneration; Blindness, Cortical; Scotoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Condition 1 - 'Scotoma awareness' Training (Experimental): Participants will be asked to report the emotion of an emoji face ('happy' vs 'sad') that could appear anywhere on screen. For the entire duration of the training, an explicit, sharp outlined occluder surrounding the participant's true retinal scotoma will be rendered on screen. This occluder will be generated through a gaze-contingent display. The size and the contrast of the target will change adaptively in response to the patient's performance.
  Interventions: Behavioral: 'Scotoma awareness' Training
- Condition 2 - Control Training (Experimental): In the control condition, participants will perform the same task as the scotoma awareness training, without the artificial visible scotoma.
  Interventions: Behavioral: Control Training

INTERVENTIONS:
Behavioral: 'Scotoma awareness' Training — In the 'scotoma awareness' training, patients will perform visual search and orientation discrimination tasks while an opaque occluder, custom-tailored to overlap each patient's retinal scotoma, is constantly presented on the computer screen.
  Arms: Condition 1 - 'Scotoma awareness' Training
Behavioral: Control Training — The task will be performed in the control group without the visible scotoma.
  Arms: Condition 2 - Control Training

SUMMARY:
The proposed research is relevant to public health because a greater understanding of plasticity after central vision loss can inform new therapies for treating low vision and has potential to benefit millions of individuals suffering from low vision. The treatment of low vision is particularly relevant to the mission of the NEI to support research on visual disorders, mechanisms of visual function and preservation of sight.

Declines in vision are particularly common in older adults and thus increasing our understanding of how to cre- ate effective means of improving vision is also highly relevant to the mission of the NIA to support research on aging and the health and well-being of older people.

DETAILED DESCRIPTION:
This proposal tests a novel 'scotoma awareness' approach to aid those with Macular Degeneration (MD). MD is the leading cause of central vision loss worldwide. MD patients spontaneously develop oculomotor strategies to overcome loss of central vision, such as developing a new peripheral fixation spot to replace the fovea (preferred retinal locus, or PRL). However, development of a PRL and the rate of success in developing one vary greatly, meaning some patients live years without making effective use of their spared vision. Recent, studies in Vision Science show that training healthy participants with gaze-contingent displays, obstructing central vision ('simulated scotoma'), leads to development of PRLs at a faster time scale than found for MD patients. Additionally, oculomotor metrics developed in our lab, are effective in characterizing individual eye movement patterns in simulated scotoma participants. The ability to describe differences in compensatory strategies in MD represents a crucial step towards individualized rehabilitative strategies, which could be further improved by accelerating PRL development. However, it is unclear whether these results can be reproduced in those with MD. It has been suggested that the visible, sharp-edged occluder in the gaze- contingent displays increases scotoma awareness, thus accelerating PRL development. Many MD patients are unaware of the location of their scotoma, with some persisting to use their damaged fovea as a fixation spot. No study to date has translated the use of a simulated scotoma to promote rapid PRL development in MD patients. As a first step towards addressing individual differences in patients and examine whether Vision Science paradigms can be used as a rehabilitative tool in MD, we propose two Aims: In Aim 1 we will use a set of oculomotor metrics to characterize individual profiles of compensation. In Aim 2 we will test the effectiveness of the visible, simulated scotoma as a technique to promote the rapid development of a PRL. Patients will undergo a 'scotoma awareness' training, in which a simulated scotoma, individually tailored for each patient, will be used to help them visualize their region of vision loss. Patients will be tested on the same metrics from Aim 1 and a battery of visual and cognitive assessments before and after the 'scotoma awareness' (or control) sessions. This will enable quantification of the effect of scotoma awareness both in terms of visual abilities and oculomotor strategies, and test the hypothesis that awareness of the location and extent of retinal damage promotes fast PRL development. While challenging, the use of eye tracking techniques in patients could be highly rewarding if this scotoma awareness procedure proves to be effective. A null result would be equally informative, suggesting fundamental differences between physiological and simulated scotomas, thus providing a limit in the use of simulations of retinal damage as a framework for the study of retinal pathologies such as MD. This will provide a unique data set to help those developing interventions for central vision loss understand how approaches to visual rehabilitation, and individual differences, give rise to training outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Severely impaired vision in both eyes (20/100 or worse)
* Diagnosis of Macular Degeneration
* Light sensitivity in the macular retina that is at least 10 dB units worse than in peripheral regions, as demonstrated by a scanning laser ophthalmoscope (SLO, MAIA)
* Medical record review indicates this disease severity level has been present for at least 2 years.

Exclusion Criteria:

* Inability to sit still in eye tracker for extended periods
* Inability to visualize iris on video eye tracker
* Bilateral retinal scotomas larger than 20° diameter

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Visual Acuity after completion of Training at approximately 6 weeks and 14 weeks | Baseline, after training completion, training is complete 6 weeks from baseline on average, and at follow up, 14 weeks from baseline on average
  Score measured on EDTRS chart
Change from Baseline Fixation stability after completion of Training at approximately 6 weeks and 14 weeks | Baseline, after training completion, training is complete 6 weeks from baseline on average, and at follow up, 14 weeks from baseline on average
  Dispersion of fixation locations averaged across trials for the PRL (expressed as the Bivariate contour ellipse area (BCEA) of the dispersion).
Change from Baseline Saccadic re-referencing after completion of Training at approximately 6 weeks and 14 weeks | Baseline, after training completion, training is complete 6 weeks from baseline on average, and at follow up, 14 weeks from baseline on average
  Proportion of trials with first fixation using PRL (expressed as a % of the total number of trials).

SECONDARY OUTCOMES:
Change from Baseline First saccade landing dispersion after completion of Training at approximately 6 weeks and 14 weeks | Baseline, after training completion, training is complete 6 weeks from baseline on average, and at follow up, 14 weeks from baseline on average
  The dispersion of the end point of the first saccade (expressed as the BCEA of the dispersion).
Change from Baseline Latency of target acquisition after completion of Training at approximately 6 weeks and 14 weeks | Baseline, after training completion, training is complete 6 weeks from baseline on average, and at follow up, 14 weeks from baseline on average
  The mean time until target is visible outside scotoma (expressed in seconds).
Change from Baseline Saccadic precision after completion of Training at approximately 6 weeks and 14 weeks | Baseline, after training completion, training is complete 6 weeks from baseline on average, and at follow up, 14 weeks from baseline on average
  The dispersion of the end point of the saccade that puts the target outside scotoma (expressed as the BCEA of the dispersion).
Change from Baseline Percentage of trials that are useful after completion of Training at approximately 6 weeks and 14 weeks | Baseline, after training completion, training is complete 6 weeks from baseline on average, and at follow up, 14 weeks from baseline on average
  How often participants place the target outside of the scotoma (% of dots in Saccadic precision relative to total trials).
Change from Baseline Minimal print size from MNREAD task after completion of Training at approximately 6 weeks and 14 weeks | Baseline, after training completion, training is complete 6 weeks from baseline on average, and at follow up, 14 weeks from baseline on average
  For the MNREAD test we will primarily rely upon minimal print size (a secondary measure of acuity)
Change from Baseline time-to-complete Trailmaking B subtest after completion of Training at approximately 6 weeks and 14 weeks | Baseline, after training completion, training is complete 6 weeks from baseline on average, and at follow up, 14 weeks from baseline on average
  We will look at time-to-complete the Trail Making B subtest, measured in seconds
Change from Baseline Contrast Sensitivity after completion of Training at approximately 6 weeks and 14 weeks | Baseline, after training completion, training is complete 6 weeks from baseline on average, and at follow up, 14 weeks from baseline on average
  Measured via Robson-Pelli charts

CONTACTS AND LOCATIONS:
Locations (1):
- UAB, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Results of the project will be submitted to the relevant repository (ClinicalTrials.gov, or Open-Science Framework) within one year of the final participant completing data collection. We expect to report participant flow by group (intervention or control), participant demographics and other baseline characteristics, outcome measures and statistical analyses, adverse events (if applicable), and limitations or caveats of our results. We also will ensure that the final protocol and statistical analysis plan are uploaded to the record.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Results of the project will be submitted to the relevant repository (ClinicalTrials.gov, or Open-Science Framework) within one year of the final participant completing data collection.